CLINICAL TRIAL: NCT03634033
Title: Statewide Implementation of CAPABLE-Community Aging in Place, Advancing Better Living for Elders in the Michigan Medicaid Home and Community Based Waiver Program
Brief Title: Implementation of CAPABLE in the Michigan Medicaid Waiver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Collaborators: Michigan State University (Other); University of Oklahoma (Other); National Institute on Aging (NIA) (NIH); Michigan Department of Health and Human Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R15AG058193-01 (NIH); R15AG058193-01A1S1 (NIH)
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Independent Living
Keywords: Implementation Science; Adoption; Sustainability; Alzheimers Disease; Dementia; CAPABLE; Randomized Controlled Trial; Intervention; Feasibility; Acceptability
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — CAPABLE protocol

STUDY DESIGN:
Intervention Model Description: Main Study: Randomized 2-Arms. Administrative Supplement: Cohort (Pilot) Study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MiCAP with IF (Main Study) (Experimental): MiCAP with Internal Facilitation will receive MiCAP (implementation strategies). Internal facilitators will be waiver site clinicians with exemplary clinical practice and/or supervisory experience, who are expected to be early adopters of CAPABLE; and will be selected by their supervisors.
  Interventions: Behavioral: MiCAP with IF (Main Study); Behavioral: MiCAP with IF and Caregiver Engagement (Administrative Supplement)
- MiCAP with IF and EF (Main Study) (Experimental): MiCAP with Internal Facilitation and External Facilitation will receive MiCAP (implementation strategies) and the addition of external facilitation. The external facilitators will be Super-Champion waiver program site clinicians from prior work who were trained and early adopters of CAPABLE; and will be selected by the research team to perform external facilitation.
  Interventions: Behavioral: MiCAP with IF (Main Study); Behavioral: MiCAP with IF and EF (Main Study)

INTERVENTIONS:
Behavioral: MiCAP with IF (Main Study) — Sites will conduct MiCAP strategies described as follows. Relationship Building; Assess readiness to implement of the site; Internal Facilitator (IF) Champion Coalition Building, which will include IFs training in CAPABLE and facilitation and online IF coalition meetings; Facilitation by the IF, which will include training the clinicians, reviewing home visits with the clinician to assure CAPABLE was provided; IF developing a clinical team for implementation of CAPABLE and leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care.
  CAPABLE is a multi-component intervention used to enhance older adults ability to function at home independently.
  Other Names: CAPABLE
Behavioral: MiCAP with IF and EF (Main Study) — Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted by External Facilitators. External Facilitators will train in facilitation. The work of the External Facilitators will be tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
  CAPABLE is a multi-component intervention used to enhance older adults ability to function at home independently.
  Other Names: CAPABLE
  Arms: MiCAP with IF and EF (Main Study)
Behavioral: MiCAP with IF and Caregiver Engagement (Administrative Supplement) — A pilot study to examine use of informal caregiver engagement to provide CAPABLE to beneficiaries with Alzheimer's Disease or other Dementia using MiCAP with Internal Facilitation (implementation strategies from the (Main Study). External facilitator will be Champion, clinician, and an early adopters of CAPABLE.
  Arms: MiCAP with IF (Main Study)

SUMMARY:
Main study: Nearly half of older adults report problems with function, which can lead to difficulty with activities of daily living and nursing home placement. Thus, there is a need to implement evidence-based models of care to improve function and those factors that support function in older adults living in the community. One such model is CAPABLE (Community Aging in Place Advancing Better Living for Elders), a person-centered, nurse and occupational therapy intervention supported by assistive devices and home modifications. The investigators build on prior work that translated CAPABLE and conducted preliminary testing of a package of implementation strategies. This R15 application will test site-level adoption and sustainability after deploying a package of implementation strategies (readiness assessment, training, facilitation, champions, coalition building, and audit and feedback). Sites will be randomized to internal facilitation alone or internal facilitation plus external facilitation. This work will impact implementation science by testing two approaches to implementation of an evidence-based intervention to improve outcomes among older adults in a Medicaid Waiver program.

ADMINISTRATIVE SUPPLEMENT We extend the Parent Trial by addressing a problem found while deploying CAPABLE with beneficiaries with Alzheimer's disease (AD) or dementia. There are 39.8 million informal caregivers in the US and 16.3 million who care for someone with AD or dementia; and 1,500 of those are in the Michigan waiver. Most beneficiaries with those conditions did not accept CAPABLE as they were unable to receive instruction. Interventions that improve caregiver knowledge, confidence, and self-efficacy improve care they provide. Thus, the goal is to extend provision of CAPABLE to beneficiaries with AD or dementia via the engagement of their informal caregivers. This work is significant as there are 1,500 beneficiaries with AD or dementia in the waiver who could benefit from CAPABLE yet many did not, as they were to receive instructions. To date, CAPABLE has only been designed to be used directly with the individuals without caregiver involvement. In the waiver, beneficiaries are required to have a designated caregiver, therefore, modifying the toolkit for use by caregivers could aid in deploying CAPABLE to beneficiaries with AD or dementia.

DETAILED DESCRIPTION:
Main study: The National Institutes of Health (NIH) defines Implementation Science (IS) as the process of applying evidence to the treatment or prevention of human disease. In response, this trial is significant because it addresses testing of multimodal implementation strategies of an evidence-based intervention (CAPABLE) in a Medicaid setting to improve the quality and effectiveness of a waiver. Investigators will utilize implementation strategies refined in prior work (MiCAP; Hartford/Hillman/CMS) where the investigators trained clinicians (N=34) and provided CAPABLE for beneficiaries (N=270).

For this application, the investigators extend their work and train "all" Registered Nurses (RNs), Occupational Therapists (OTs), and Social Workers (SWs) (N=575) in the waiver sites in Michigan to implement the CAPABLE model of care for "all" Medicaid waiver beneficiaries (N=15,000). Guided by site managers, the team will select and train Internal Facilitators (IFs), who are supervisors/employees that work for the waiver site, to conduct facilitation at each site as "Champions". Investigators will utilize waiver employees as External Facilitators (EFs), who were early adopters of CAPABLE in prior work, as "Super-Champions" for Arm 2.

This trial is also significant as it addresses a critical barrier to implementation of evidence-based interventions to improve function in older adults living in the community to age-in-place (CAPABLE). Evidence suggest 90% of older adults prefer to age-in-place; yet a gap exists between their desire and ability. Thus, further testing of efficacy of an intervention (CAPABLE) in a Medicaid waiver population will fill a gap in science and build upon evidence.

The Institute of Medicine, NIH, and the Agency for Healthcare Research and Quality have each established IS as a research priority so that the benefits of evidence-based interventions can be realized. Consequently, strategies (MiCAP) to overcome barriers and increase the pace and the effectiveness of implementation are a public health priority. The multimodal implementation strategies (MiCAP N=6) include: assessing readiness, conducting training, using IF Champions, building an IF coalition, and audit and feedback is adequate. Additionally, investigators will examine if the additive EF is required to support adoption and sustainability of an evidence-based intervention (CAPABLE).

Disabilities in basic activities of daily living (ADLs [e.g., bathing, toileting]) and instrumental ADLs (IADL [e.g., shopping, cleaning]) are the primary modifiable predictors of nursing home (NH) placement. Disability is also a major driver of increased risk of falls and may lead to poor quality-of-life. Disability creates an inability to carry out everyday ADLs. There are a number of risks for disability like complex medication regimens, poor balance and strength, inadequate communication with clinicians, falling, and unsafe ADL performance. In addition, unsafe environments and deteriorated housing increase risk.

To address this problem, the evidence-based intervention, CAPABLE, addresses modifiable intrinsic and extrinsic risk factors and considers the psychological, environmental, and physical factors to enhance function of disabled individuals and promote aging-in-place. A multi-component model of care, CAPABLE was designed to reduce the effect of problems with physical function among low-income older adults living at home by addressing an individual's capabilities and the home environment.

CAPABLE was adapted from the ABLE program. ABLE used a person-directed, consultative model involving 6 home sessions conducted by OTs and physical therapists who provided home alterations (assistive devices [e.g., shower chair, reacher, raised toilet seat], environmental modifications [e.g., grab bar, ramps], and select home modifications [e.g., widen bathroom doorway]) and instruction in various techniques to enable participants to achieve self-identified functional goals. CAPABLE is a 16-week structured program delivered by OTs who conduct 6 home visits and provide assistive devices, RNs who conduct 4 home visits, and a repairperson who provides home alterations (i.e., installs devices, environmental modifications, and home repair). CAPABLE's interdisciplinary team provides consultation with older adults to help them identify daily activity goals (e.g., taking a shower, walking to the bathroom), evaluate barriers to achieving those goals, and attain outcomes collaboratively. The OT addresses ADLs, IADLs, and discretionary activities at home such as functional mobility, meal preparation, bathing, and dressing. The RN targets underlying issues that influence ADLs, IADLs, and discretionary activities at home, such as pain reduction, improvement in mood, fall prevention, medication review and management, primary care physician communication, incontinence management, sexual health, and smoking cessation. CAPABLE draws upon approaches to enhance uptake and adoption of strategies by patients by assessing readiness and using motivational interviewing.

In this trial, the investigators move IS forward by examining a multimodal implementation strategy (MiCAP) approach to implement evidence (CAPABLE) in a Medicaid Waiver program. To fill an IS gap, investigators will use proven implementation strategies that are packaged (MiCAP) and delivered to clinicians in the waiver program sites to support beneficiary improvement in function and those factors that influence function in older disabled adults aging-in-place.

ADMINISTRATIVE SUPPLEMENT There is a paucity of literature on caregiver provision of assessment or direct care to individuals with AD or dementia, as most discuss burden, confidence, stress, depression, or health. In 2005, the AARP used a Delphi technique to identify caregiver competency domains of medical/nursing skills, assessment, measurement, collaborating, and communication. A review of caregiver training programs found problem solving, use of community resources, and communication to be the primary focus. Physical or emotional assessment, medical/nursing skills training, home exercises, medication management, or planning, like what is needed when delivering CAPABLE, appeared to be lacking in caregiver training. Regarding toolkit usage, Powell and colleagues recommend using toolkits when implementing interventions, and our parent trial uses a beneficiary toolkit. A recent review of 72 studies evaluating use of toolkits (i.e. weight management, fall prevention, vaccination, pain management, and patient safety) found 57% reported adherence to clinical procedures and toolkit effects were positive. This finding supports use of a toolkit with caregivers when CAPABLE is deployed with beneficiaries with AD or dementia. Many older adults cared for by informal caregivers have unmet needs. A 44.3% (38.2% ADL related, 14.6% IADL related) unmet need rate is common among older adults with caregivers. Higher rates of unmet needs are likely in beneficiaries in the waiver as they are multi-morbid and low-income with few resources and even worse in those with AD or dementia.

ELIGIBILITY:
MAIN TRIAL:

Inclusion Criteria: Waiver program site must be under contract as a Home and Community Based Services (HCBS) waiver provider in Michigan (including clinicians and beneficiaries). Waiver program site must use the Center for Information Management (CIM) electronic health record.

Exclusion Criteria: Waiver program site not under contract as a HCBS waiver provider in Michigan. Waiver program site not using the single electronic health record from Center for Information Management (CIM).

ADMINISTRATIVE SUPPLEMENT (all in main trial plus below):

Inclusion Criteria: Caregivers designated in beneficiary's record, and beneficiary diagnosed with Alzheimer's Disease or dementia.

Exclusion Criteria: Without a caregiver or beneficiary not diagnosed with Alzheimer's Disease or dementia.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7777 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Spoelstra, PhD, Principal Investigator — Grand Valley State University
Locations (18):
- United States (18):
  - Northeast Michigan Community Service Agency (NEMCSA), Alpena, Michigan
  - Region 3B Area Agency on Aging/CareWell Services Southwest, Battle Creek, Michigan
  - Region VII Area Agency on Aging, Bay City, Michigan
  - Region 2 Area Agency on Aging, Brooklyn, Michigan
  - Macomb-Oakland Regional Center Home Care, Inc., Clinton Township, Michigan
  - Detroit Area Agency on Aging, Detroit, Michigan
  - UPCAP, Escanaba, Michigan
  - Valley Area Agency on Aging, Flint, Michigan
  - Area Agency on Aging of Western Michigan, Inc., Grand Rapids, Michigan
  - Senior Services, Kalamazoo, Michigan
  - Tri-County Office on Aging, Lansing, Michigan
  - Senior Resources, Muskegon, Michigan
  - A&D Home Health Care, Inc., Saginaw, Michigan
  - Region IV Area Agency on Aging, Saint Joseph, Michigan
  - The Information Center, Taylor, Michigan
  - Northern Lakes Community Mental Health/Northern Health Care Management, Traverse City, Michigan
  - Area Agency on Aging of Northwest Michigan, Traverse City, Michigan
  - The Senior Alliance, Wayne, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spoelstra SL, Schueller M, Sikorskii A. Testing an implementation strategy bundle on adoption and sustainability of evidence to optimize physical function in community-dwelling disabled and older adults in a Medicaid waiver: a multi-site pragmatic hybrid type III protocol. Implement Sci. 2019 Jun 13;14(1):60. doi: 10.1186/s13012-019-0907-1. PMID 31196137
- [Result] Spoelstra SL, Schueller M, Dorn E, Sikorskii A. Measuring Organizational Readiness for Change in Michigan's Home and Community-based Services Program: Instrument Adaptation and Psychometric Testing. Home Health Care Serv Q. 2022 Jul-Sep;41(3):255-266. doi: 10.1080/01621424.2022.2077161. Epub 2022 May 18. PMID 35585762
- [Derived] Spoelstra SL, Schueller M, Basso V, Sikorskii A. Results of a multi-site pragmatic hybrid type 3 cluster randomized trial comparing level of facilitation while implementing an intervention in community-dwelling disabled and older adults in a Medicaid waiver. Implement Sci. 2022 Aug 26;17(1):57. doi: 10.1186/s13012-022-01232-5. PMID 36028873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: MAIN STUDY. Group allocation-randomized 18 waiver sites, 9 to MiCAP with IF; and 9 to MiCAP with IF and EF. Recruited 2 groups of participants at each site: clinicians employed by the sites to provide the intervention to waiver beneficiaries to receive the intervention.
  ADMINISTRATIVE SUPP. No group allocation: Recruited 3 groups of participants at 3 sites from Main Study; clinicians employed at sites, caregivers to provide the intervention, and beneficiaries to receive it; plus MiCAP IF.
Pre-assignment Details: COUNT OF PARTICIPANTS: for ARMS/GROUPS- Some clinicians/beneficiaries in MiCAP with IF Main Study may be represented in Administrative Supplement: clinicians/beneficiaries; counted more than once/signed more than 1 Consent Form.
  MAIN STUDY: UNITS- MiCAP with IF/IF+EF Beneficiaries and Clinicians use the same 18 sites.
  ADMINISTRATIVE SUPPLEMENT: Some caregivers dropped out of study after beneficiary passed away or transferred to a facility; the caregiver was not deceased or in a facility.
Units Other Than Participants: Sites (Main Study only)
Groups:
- MiCAP With IF (Main Study: Beneficiaries); MiCAP With IF (Main Study: Clinicians): MiCAP with Internal Facilitation will receive MiCAP (implementation strategies). Internal facilitators will be waiver site clinicians with exemplary clinical practice and/or supervisory experience, who are expected to be early adopters of CAPABLE; and will be selected by their supervisors.
  MiCAP with IF: Sites will conduct MiCAP strategies described as follows. Relationship Building; Assess readiness to implement of the site; Internal Facilitator (IF) Champion Coalition Building, which will include IFs training in CAPABLE and facilitation and online IF coalition meetings; Facilitation by the IF, which will include training the clinicians, reviewing home visits with the clinician to assure CAPABLE was provided; IF developing a clinical team for implementation of CAPABLE and leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care
- MiCAP With IF and EF (Main Study: Beneficiaries); MiCAP With IF and EF (Main Study: Clinicians): MiCAP with Internal Facilitation and External Facilitation will receive MiCAP (implementation strategies) and the addition of external facilitation. The external facilitators will be Super-Champion waiver program site clinicians from prior work who were trained and early adopters of CAPABLE; and will be selected by the research team to perform external facilitation.
  MiCAP with IF and EF: Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted by External Facilitators. External Facilitators will train in facilitation. The work of the External Facilitators will be tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
- Administrative Supplement: Clinicians: Clinicians who were employed at the waiver sites and were trained in using CAPABLE with caregivers of beneficiaries with Alzheimer's Disease or Dementia; plus MiCAP with IF from Main Study.
- Administrative Supplement: Caregivers: Caregivers of beneficiaries diagnosed with Alzheimer's Disease or Dementia who agreed to assist with providing CAPABLE to their beneficiary; plus MiCAP with IF from Main Study.
- Administrative Supplement: Beneficiaries: Beneficiaries enrolled at the waiver who were diagnosed with Alzheimer's Disease or Dementia and needed to receive CAPABLE; ; plus MiCAP with IF from Main Study.
Period: Overall Study
Arm/Group | MiCAP With IF (Main Study: Beneficiaries) | MiCAP With IF and EF (Main Study: Beneficiaries) | MiCAP With IF (Main Study: Clinicians) | MiCAP With IF and EF (Main Study: Clinicians) | Administrative Supplement: Clinicians | Administrative Supplement: Caregivers | Administrative Supplement: Beneficiaries
Started | 3497; 9 Sites (Main Study only) | 3533; 9 Sites (Main Study only) | 282; 9 Sites (Main Study only) | 257; 9 Sites (Main Study only) | 106; 3 Sites (Main Study only) | 50; 3 Sites (Main Study only) | 52; 3 Sites (Main Study only)
Completed | 3113; 9 Sites (Main Study only) | 3242; 9 Sites (Main Study only) | 168; 9 Sites (Main Study only) | 96; 9 Sites (Main Study only) | 101; 3 Sites (Main Study only) | 37; 3 Sites (Main Study only) | 37; 3 Sites (Main Study only)
Not Completed | 384; 0 Sites (Main Study only) | 291; 0 Sites (Main Study only) | 114; 0 Sites (Main Study only) | 161; 0 Sites (Main Study only) | 5; 0 Sites (Main Study only) | 13; 0 Sites (Main Study only) | 15; 0 Sites (Main Study only)
Not completed — Did not have a post-assessment | 384 | 291 | 114 | 161 | 5 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 7 | 7
Not completed — In Assisted Living/Nursing Home/Hospice | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Main Study: MiCAP With IF (Beneficiaries); Main Study: MiCAP With IF (Clinicians): MiCAP with Internal Facilitation will receive MiCAP (implementation strategies). Internal facilitators will be waiver site clinicians with exemplary clinical practice and/or supervisory experience, who are expected to be early adopters of CAPABLE; and will be selected by their supervisors.
  MiCAP with IF: Sites will conduct MiCAP strategies described as follows. Relationship Building; Assess readiness to implement of the site; Internal Facilitator (IF) Champion Coalition Building, which will include IFs training in CAPABLE and facilitation and online IF coalition meetings; Facilitation by the IF, which will include training the clinicians, reviewing home visits with the clinician to assure CAPABLE was provided; IF developing a clinical team for implementation of CAPABLE and leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care
- Main Study: MiCAP With IF+EF (Beneficiaries); Main Study: MiCAP With IF+EF (Clinicians): MiCAP with Internal Facilitation and External Facilitation will receive MiCAP (implementation strategies) and the addition of external facilitation. The external facilitators will be Super-Champion waiver program site clinicians from prior work who were trained and early adopters of CAPABLE; and will be selected by the research team to perform external facilitation.
  MiCAP with IF and EF: Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted by External Facilitators. External Facilitators will train in facilitation. The work of the External Facilitators will be tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
- Administrative Supplement: Clinicians: Clinicians who were employed at the waiver sites and were trained in using the toolkit when implementing CAPABLE with caregivers of beneficiaries with Alzheimer's Disease or Dementia.
- Administrative Supplement: Caregivers: Caregivers of beneficiaries diagnosed with Alzheimer's Disease or Dementia who will receive the toolkit to assist in taking care of their beneficiary.
- Administrative Supplement: Beneficiaries: Beneficiaries enrolled at the waiver who were diagnosed with Alzheimer's Disease or Dementia.
- Total: Total of all reporting groups
Arm/Group | Main Study: MiCAP With IF (Beneficiaries) | Main Study: MiCAP With IF+EF (Beneficiaries) | Main Study: MiCAP With IF (Clinicians) | Main Study: MiCAP With IF+EF (Clinicians) | Administrative Supplement: Clinicians | Administrative Supplement: Caregivers | Administrative Supplement: Beneficiaries | Total
Number analyzed (Participants) | 3497 | 3533 | 282 | 257 | 106 | 50 | 52 | 7777
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (14.58) | 71.19 (14.02) | 43.07 (11.57) | 47.00 (11.59) | 45.78 (10.48) | 63.28 (11.29) | 81.23 (9.27) | 70.35 (14.32)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 1137 | 1130 | 16 | 22 | 3 | 10 | 12 | 2330
  Sex: Female | 2360 | 2403 | 266 | 231 | 103 | 40 | 40 | 5443
  Sex: Unknown | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 108 | 97 | 13 | 5 | 5 | 1 | 1 | 230
  Not Hispanic or Latino | 3357 | 3401 | 267 | 247 | 101 | 49 | 51 | 7473
  Unknown or Not Reported | 32 | 35 | 2 | 5 | 0 | 0 | 0 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 25 | 9 | 5 | 1 | 0 | 1 | 1 | 42
  Asian | 25 | 25 | 1 | 4 | 0 | 0 | 1 | 56
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 7
  Black or African American | 541 | 1228 | 14 | 39 | 2 | 4 | 4 | 1832
  White | 2735 | 2122 | 248 | 202 | 99 | 44 | 46 | 5496
  More than one race | 49 | 33 | 10 | 4 | 0 | 1 | 0 | 97
  Unknown or Not Reported | 119 | 112 | 4 | 7 | 5 | 0 | 0 | 247
Region of Enrollment [Number; unit: participants]
  United States | 3497 | 3533 | 282 | 257 | 106 | 50 | 52 | 7777
Emergency Department Visits [Number; unit: Number on scale] — Population: ED data was not collected for MiCAP with IF (Main Study: Clinicians), MiCAP with IF and EF (Main Study: Clinicians), Administrative Supplement: Clinicians, and Administrative Supplement: Caregivers.
  Number on scale
    number analyzed (Participants) | 3497 | 3533 | 0 | 0 | 0 | 0 | 52 | 7082
    (all) | 450 | 421 |  |  |  |  | 12 | 883

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Effect of MiCAP With IF Alone Versus MiCAP With IF+EF on Site-level Outcomes of Adoption and Sustainability of CAPABLE
Description: Adoptions and sustainability of the intervention using the Stages of Implementation Completion (SIC) at a site (18). SIC is a tool that tracks achievement of key activities when implementing an evidence-based intervention.
  SIC has 6 stages with multiple implementation activities; each activity had an assigned numeric value and when a activity was completed, a score was assigned. The *total* SIC score ranges from 0-100. Stage 1 score range 0-12. Stage 2 0-16. Stage 3 0-24. Stage 4 0-16. Stage 5 0-16. Stage 6 0-16. The *total* score was calculated by summing the points of each stage. The higher the *total* score, the more implementation activities were completed.
  For the below reported *total* score, each waiver site had their *total* SIC score numerically calculated. Then, the mean and standard deviation were calculated by group/arm.
Time Frame: 9 months
Population: The participants analyzed were the 18 waiver sites from the MAIN STUDY that were then randomized to either MiCAP with IF (n=9) or MiCAP with IF and EF (n=9).
  The Administrative Supplement Arms/Groups are not included in this outcome as data were only collected during the main study.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: waiver sites
Groups:
- MiCAP With IF: MiCAP with Internal Facilitation will receive MiCAP (implementation strategies). Internal facilitators will be waiver site clinicians with exemplary clinical practice and/or supervisory experience, who are expected to be early adopters of CAPABLE; and will be selected by their supervisors.
  MiCAP with IF: Sites will conduct MiCAP strategies described as follows. Relationship Building; Assess readiness to implement of the site; Internal Facilitator (IF) Champion Coalition Building, which will include IFs training in CAPABLE and facilitation and online IF coalition meetings; Facilitation by the IF, which will include training the clinicians, reviewing home visits with the clinician to assure CAPABLE was provided; IF developing a clinical team for implementation of CAPABLE and leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care
- MiCAP With IF and EF: MiCAP with Internal Facilitation and External Facilitation will receive MiCAP (implementation strategies) and the addition of external facilitation. The external facilitators will be Super-Champion waiver program site clinicians from prior work who were trained and early adopters of CAPABLE; and will be selected by the research team to perform external facilitation.
  MiCAP with IF and EF: Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted by External Facilitators. External Facilitators will train in facilitation. The work of the External Facilitators will be tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
Arm/Group | MiCAP With IF | MiCAP With IF and EF
Number analyzed (Participants) | 3779 | 3790
Number analyzed (waiver sites) | 9 | 9
score on a scale | 72.22 (16.98) | 61.33 (19.29)
Statistical Analysis 1: Comparison: MiCAP With IF vs MiCAP With IF and EF; Given 18 sites (9 in each arm) available in Michigan, in the comparison of site-level outcome of adoption and sustainability, the detectable effect size with power of 0.80 in two-sided tests at .05 level of significance was d=1.41; Test type: Superiority — Examination of intensity of facilitation (IF vs IF+EF) on adoption and sustainability using an evidence-based intervention (CAPABLE); p = 0.22, t-test, 2 sided — A priori threshold for statistical significance was .05; 16 degrees of freedom for the t-test comparing two independent groups, n=9 each; Mean Difference (Final Values) = 10.89, 95% CI 2-sided [-7.27 to 29.05], Standard Deviation 18.17

2. Secondary Outcome: Main Study: Beneficiary's ADLs Summed Score
Description: Activities of Daily Living (ADLs) data were collected from the Minimum Data Set-Home Care (MDS-HC) in the Electronic Health Record (EHR). MDS-HC is a person-centered assessment for the collection of minimum essential nursing data, with reliability and validity, and used in the Michigan Medicaid Waiver program.
  The score is a summed score of 11 items on the MDS-HC; with a score range of 0-88. The lower the summed score, the more independent the beneficiary is at performing ADLs. For the 11 items, the available scores are 0= Independent, 1= Set-up help only, 2= Supervision, 3= Limited assistance, 4= Extensive assistance, 5= Maximal assistance, 6= Total dependence, 8= Activity did not occur during entire period.
Time Frame: Exit (9-months)
Population: Participants analyzed were the beneficiaries at sites (18); arms included randomized to either MiCAP with IF (n=9) or MiCAP with IF and EF (n=9).
Measure: Mean (Standard Error); unit: Score on scale
Units Other Than Participants: Waiver Sites
Arm/Group | MiCAP With IF (Main Study: Beneficiaries) | MiCAP With IF and EF (Main Study: Beneficiaries)
Number analyzed (Participants) | 3113 | 3242
Number analyzed (Waiver Sites) | 9 | 9
Score on scale | 26.13 (0.20) | 25.85 (0.19)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Study: Beneficiaries) vs MiCAP With IF and EF (Main Study: Beneficiaries); Adjusted means at month 9 were calculated adjusting for baseline value of the outcome and nesting of participants within sites; Test type: Superiority — Examination of intensity of facilitation (IF vs IF+EF) on beneficiaries ADLs at exit using an evidence-based intervention (CAPABLE); p = 0.73, Mixed Models Analysis — A priori threshold for statistical significance was .05; no adjustments for multiple comparisons; F-test was used built into mixed models that adjusted for clustering via a random effect of site; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.16 to 0.73], Standard Error of Mean 0.23 — IF minus IF+EF

3. Secondary Outcome: Main Study: Beneficiary's IADLs
Description: Instrumental Activities of Daily Living (IADLs) was collected from the Minimum Data Set-Home Care (MDS-HC) in the Electronic Health Record (EHR). MDS-HC is a person-centered assessment for the collection of minimum essential nursing data, with reliability and validity, and used in the Michigan Medicaid Waiver program.
  The below reported score is a summed score of 8 items on the MDS-HC; summed score range is 0-64. The lower the summed score, the more independent the beneficiary is at performing IADLs. For the 8 items, the available scores are 0= Independent, 1= Set-up help only, 2= Supervision, 3= Limited assistance, 4= Extensive assistance, 5= Maximal assistance, 6= Total dependence, 8= Activity did not occur during entire period.
Time Frame: Exit (9-months)
Population: The participants analyzed were the 18 waiver sites from the MAIN STUDY that were then randomized to either MiCAP with IF (n=9) or MiCAP with IF and EF (n=9).
  Arms /Groups MiCAP with IF (Main Study: Clinicians), MiCAP with IF and EF (Main Study: Clinicians), Administrative Supplement: Clinicians, and Administrative Supplement: Caregivers, and Administrative Supplement: Beneficiaries were not included as data was not collected.
Measure: Mean (Standard Error); unit: Score on scale
Units Other Than Participants: Waiver Sites
Arm/Group | MiCAP With IF (Main Study: Beneficiaries) | MiCAP With IF and EF (Main Study: Beneficiaries)
Number analyzed (Participants) | 3113 | 3242
Number analyzed (Waiver Sites) | 9 | 9
Score on scale | 29.54 (0.17) | 29.24 (0.17)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Study: Beneficiaries) vs MiCAP With IF and EF (Main Study: Beneficiaries); Post-intervention means were compared adjusting for baseline values and nesting of participants within sites; Test type: Superiority — Examination of intensity of facilitation (IF vs IF+EF) needed on beneficiaries IADLs using an evidence-based intervention (CAPABLE); p = 0.15, Mixed Models Analysis — Threshold for statistical significance was .05 with no adjustments for multiple comparisons; F-test was used built into mixed models that adjusted for clustering; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.11 to 0.72], Standard Error of Mean 0.21 — IF minus IF+EF

4. Secondary Outcome: Main Study: Beneficiary's Pain
Description: Pain data were collected from the Minimum Data Set-Home Care (MDS-HC) in the Electronic Health Record (EHR). MDS-HC is a person-centered assessment for the collection of minimum essential nursing data, with reliability and validity, and used in the Michigan Medicaid Waiver program.
  The score is a summed score of 4 self-reported items on the MDS-HC; the summed score range is 0-11. The lower the summed score, the less pain the beneficiary reported. The four items included: pain frequency (range 0-3); pain intensity (0-4); pain consistency (0-3); and breakthrough pain (0-1).
Time Frame: Exit (9-months)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on scale
Units Other Than Participants: Waiver Sites
Arm/Group | MiCAP With IF (Main Study: Beneficiaries) | MiCAP With IF and EF (Main Study: Beneficiaries)
Number analyzed (Participants) | 3113 | 3242
Number analyzed (Waiver Sites) | 9 | 9
Score on scale | 7.52 (0.13) | 7.44 (0.13)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Study: Beneficiaries) vs MiCAP With IF and EF (Main Study: Beneficiaries); Test type: Superiority — Examination of intensity of facilitation (IF vs IF+EF) needed on beneficiaries pain at exit using an evidence-based intervention (CAPABLE); p = 0.61, Mixed Models Analysis — Threshold for statistical significance was.05; no adjustments for multiple comparisons; F-test was used built into mixed models that adjusted for clustering; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.23 to 0.39], Standard Error of Mean 0.16 — IF minus IF+EF

5. Secondary Outcome: Main Study: Beneficiary's Depression
Description: Depression was collected from the Minimum Data Set-Home Care (MDS-HC) in the Electronic Health Record (EHR). MDS-HC is a person-centered assessment for the collection of minimum essential nursing data, with reliability and validity, and used in the Michigan Medicaid Waiver program.
  The below reported score is a summed score of 3 self-reported items on the MDS-HC; the summed score range is 0-24. The lower the summed score, the less depressed the beneficiary reported. The 3 items included: little interest in things; anxious, restless, or uneasy; and sad, depressed, or hopeless. For the 3 items, the available scores are 0= Not in last 3 days, 1= Not in last 3 days, but often feels that way, 2= In 1-2 days of last 3 days, 3= Daily in last 3 days, 8= Person could not (would not) respond.
Time Frame: Exit (9-months)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on scale
Units Other Than Participants: Waiver Sites
Arm/Group | MiCAP With IF (Main Study: Beneficiaries) | MiCAP With IF and EF (Main Study: Beneficiaries)
Number analyzed (Participants) | 3113 | 3242
Number analyzed (Waiver Sites) | 9 | 9
Score on scale | 1.3 (0.05) | 1.17 (0.05)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Study: Beneficiaries) vs MiCAP With IF and EF (Main Study: Beneficiaries); Test type: Superiority — Examination of intensity of facilitation (IF vs IF+EF) needed on beneficiaries depression (baseline to exit) using an evidence-based intervention (CAPABLE); p = 0.04, F-test; F-test was used (related to the t-test arithmetically), built into mixed models that adjusted for clustering; LS Means = 0.05, 95% CI 2-sided [0.01 to 0.24], Standard Error of Mean 0.05

6. Secondary Outcome: Main Study: Beneficiary's Fall Rate
Description: Beneficiary falls data were collected from the Minimum Data Set-Home Care (MDS-HC) in the Electronic Health Record. MDS-HC is a person-centered assessment for the collection of minimum essential nursing data, with reliability and validity, and used in the Michigan Medicaid Waiver program.
  Falls were reported as proportions of occurrences on the MDS-HC; and calculated for this study based on the occurrence of a fall where yes=1 and no=0 divided by the number of participants.
Time Frame: Exit (9-months)
Measure: Mean (Standard Error); unit: percentage of participants
Groups:
- MiCAP With IF (Main Trial): MiCAP with Internal Facilitation will receive MiCAP (implementation strategies). Internal facilitators will be waiver site clinicians with exemplary clinical practice and/or supervisory experience, who are expected to be early adopters of CAPABLE; and will be selected by their supervisors.
  MiCAP with IF (Main Trial): Sites will conduct MiCAP strategies described as follows. Relationship Building; Assess readiness to implement of the site; Internal Facilitator (IF) Champion Coalition Building, which will include IFs training in CAPABLE and facilitation and online IF coalition meetings; Facilitation by the IF, which will include training the clinicians, reviewing home visits with the clinician to assure CAPABLE was provided; IF developing a clinical team for implementation of CAPABLE and leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care
- MiCAP With IF and EF (Main Trial): MiCAP with IF and EF will receive MiCAP (implementation strategies) and the addition of external facilitation. The external facilitators will be Champion who was trained and is an adopter of CAPABLE.
  MiCAP with IF (Main Trial): Sites will conduct MiCAP strategies described. Relationship Building; Assess readiness to implement of the site; Internal Facilitator (IF) Coalition Building, which will include IFs training in CAPABLE and facilitation and IF coalition meetings; Facilitation by the IF, will include training clinicians, reviewing home visits with clinicians to assure CAPABLE was provided; developing a clinical team to implement CAPABLE and leading interdisciplinary coordination; Intervention and implementation audits provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement (Main Trial): Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
Arm/Group | MiCAP With IF (Main Trial) | MiCAP With IF and EF (Main Trial)
Number analyzed (Participants) | 3397 | 3533
percentage of participants | 0.15 (0.01) | 0.14 (0.01)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Trial) vs MiCAP With IF and EF (Main Trial); Test type: Superiority — Examination of intensity of facilitation (IF vs IF+EF) on beneficiaries fall rates at exit after an evidence-based intervention (CAPABLE); p = 0.18, Mixed Models Analysis; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.93 to 1.45], Standard Error of Mean .01
Statistical Analysis 2: Comparison: MiCAP With IF (Main Trial) vs MiCAP With IF and EF (Main Trial); Occurrence of falls was analyzed with adjustment for baseline and nesting of participants within sites; Test type: Superiority; p = .18, Mixed Models Analysis — Threshold for statistical significance was .05; no adjustment for multiple comparisons; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.93 to 1.45] — Odds ratio for IF versus IF+EF

7. Secondary Outcome: Main Study: Beneficiary's Emergency Department (ED) Visits Occurrences Out of Total Number of Participants.
Description: Beneficiary-level outcome emergency department (ED) data were collected from the Minimum Data Set-Home Care (MDS-HC) in the Electronic Health Record. MDS-HC is a person-centered assessment for the collection of minimum essential nursing data, with reliability and validity, and used in the Michigan Medicaid Waiver program.
  ED visits were reported as proportion calculated based on the occurrence of an ED visit where yes=1 and no=0 out of the number of participants.
Time Frame: Exit (9-months)
Measure: Mean (Standard Error); unit: percentage of participants
Groups:
- MiCAP With IF and EF (Main Trial): MiCAP with IF and EF will receive MiCAP (implementation strategies) and the addition of EF. EF will be a waiver program clinicians trained and early adopters of CAPABLE.
  MiCAP with IF (Main Trial): Sites will conduct MiCAP strategies. Relationship Building; Assess readiness to implement of the site; IF Coalition Building; Facilitation by the IF, which will include training the clinicians, reviewing home visits to assure CAPABLE was provided; developing a clinical team for implementation of CAPABLE; leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care
  MiCAP with IF and EF (Main Trial): Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted by External Facilitators. External Facilitators will train in facilitation. The work of the External Facilitators will be tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
Arm/Group | MiCAP With IF (Main Trial) | MiCAP With IF and EF (Main Trial)
Number analyzed (Participants) | 3387 | 3533
percentage of participants | 0.92 (.01) | 0.91 (.01)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Trial) vs MiCAP With IF and EF (Main Trial); Test type: Superiority — Examination of intensity of facilitation (IF vs IF+EF) on beneficiaries ED Visits at exit after an evidence-based intervention (CAPABLE); p = 0.86, Mixed Models Analysis — Threshold for statistical significance was .05 with no adjustments for multiple comparisons; Adjustment for baseline and nesting of participants within sites; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.79 to 1.22], Standard Error of Mean 0.01

8. Secondary Outcome: Main Study: Beneficiary's Hospitalization Occurrences Out of Total Number of Participants.
Description: Beneficiary-level outcomes hospitalizations data were collected from the Minimum Data Set-Home Care (MDS-HC) in the Electronic Health Record. MDS-HC is a person-centered assessment for the collection of minimum essential nursing data, with reliability and validity, and used in the Michigan Medicaid Waiver program.
  Hospitalizations were reported based on the occurrence and calculated for this study as rates of hospitalization where yes=1 and no=0 out of total number of participants.
Time Frame: Exit (9-months)
Measure: Mean (Standard Error); unit: percentage of participants
Groups:
- MiCAP With IF and EF (Main Trial): MiCAP with IF and EF will receive MiCAP (implementation strategies) and the addition of external facilitation. The EF will be a Champion waiver trained and an adopter of CAPABLE.
  MiCAP with IF (Main Trial): Sites will conduct MiCAP strategies. Relationship Building; Assess readiness to implement of the site; Facilitation by the IF, which will include training the clinicians, reviewing home visits with the clinician to assure CAPABLE was provided; IF developing a clinical team and leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care
  MiCAP with IF and EF (Main Trial): Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted by External Facilitators. External Facilitators will train in facilitation. The work of the External Facilitators will be tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
Arm/Group | MiCAP With IF (Main Trial) | MiCAP With IF and EF (Main Trial)
Number analyzed (Participants) | 3387 | 3553
percentage of participants | 0.01 (.01) | .01 (.01)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Trial) vs MiCAP With IF and EF (Main Trial); Test type: Superiority — Examination of intensity of facilitation (IF vs IF+EF) needed on beneficiaries hospitalizations (baseline to exit) using an evidence-based intervention (CAPABLE); p = 0.95, F-test; F-test was used (related to the t-test arithmetically), built into mixed models that adjusted for clustering; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.72 to 1.42], Standard Error of Mean 1.01

9. Other Pre Specified Outcome: Main Study: Clinician Attitude Towards Evidence Based Practice Use
Description: Evidence-Based Practice Attitude Scale (EBPAS-50) is a 50-item tool that assesses clinician attitudes toward adopting evidence into practice. EBPAS-50 has 50 items on the tool which includes 10 sub-scales: limitations, openness, monitoring, requirements, employability, feedback, burden, appeal, divergence, balance; and the questions are negatively framed. The 10 sub-scales are summed into a higher order total scale score representing respondent's attitude toward adopting evidence into practice.
  EBPAS-50 total scale score ranges from 0-200 with higher being a better attitude towards use of evidence in practice. Each of the 10 sub-scales ranges from 0-20; with higher being a better attitude towards use of evidence.
  Items are reversed scored, and the mean sub-scale scores are recomputed, before a mean score for the total EBPAS-50 item score is computed.
  A higher total score indicate a more positive attitude towards adoption of evidence-based practice use.
Time Frame: Exit (9-months)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- MiCAP With IF and EF (Main Trial): MiCAP with IF and EF will receive MiCAP (implementation strategies) and the addition of external facilitation. EF will be a Champion clinician early adopters of CAPABLE.
  MiCAP with IF (Main Trial): Sites will conduct MiCAP strategies. Relationship Building; Assess readiness to implement of the site; IF Coalition Building; Facilitation will include training clinicians, reviewing home visits to assure CAPABLE was provided; IF developing a clinical team for implementation of CAPABLE and leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care
  MiCAP with IF and EF (Main Trial): Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted by External Facilitators. External Facilitators will train in facilitation. The work of the External Facilitators will be tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
Arm/Group | MiCAP With IF (Main Trial) | MiCAP With IF and EF (Main Trial)
Number analyzed (Participants) | 282 | 257
units on a scale
  Attitude limitations | 0.00 (0.11) | -0.06 (0.11)
  Attitude openness | 0.08 (0.08) | 0.00 (0.08)
  Attitude monitoring | 0.01 (0.14) | 0.18 (0.14)
  Attitude requirements | 0.15 (0.09) | 0.18 (0.14)
  Attitude employabilty | -0.17 (0.07) | -0.04 (0.11)
  Attitude feedback (higher is better) | 0.10 (0.11) | -0.01 (0.12)
  Attitude burden | 0.13 (0.15) | 0.04 (0.14)
  Attitude appeal | 0.06 (0.08) | -0.11 (0.08)
  Attitude divergence | 0.07 (0.09) | 0.14 (0.09)
  Attitude balance | 0.11 (0.11) | 0.21 (0.10)
  Overall Attitude (total summed mean score) | -103.49 (0.92) | -103.52 (0.92)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Trial) vs MiCAP With IF and EF (Main Trial); Mixed modeling was used to account for nesting of clinicians within sites; Test type: Superiority — Examination of clinician attitude on facilitation (IF vs IF+EF) at exit when using an evidence-based intervention (CAPABLE); p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 5.11, 95% CI 2-sided [0.09 to 10.14], Standard Error of Mean 2.55

10. Other Pre Specified Outcome: Main Study: Clinician Self-efficacy
Description: General Self-efficacy (GSE) is a 10-item tool (Cronbach .79-.90) with a 4-point scale summed to 10-40, with a higher score indicating more self-efficacy.
Time Frame: Exit (9-months)
Population: Clinicians.
Measure: Mean (Standard Error); unit: Score on scale
Groups:
- MiCAP With IF and EF (Main Trial): MiCAP with IF and EF will receive MiCAP (implementation strategies) and the addition of EF. EF will be a Champion clinician and an early adopters of CAPABLE.
  MiCAP with IF (Main Trial): Sites will conduct MiCAP strategies described as follows. Relationship Building; Assess readiness to implement of the site; Champion Coalition Building; Facilitation by IF, includes training clinicians, reviewing home visits to assure CAPABLE was provided; developing a clinical team to implement CAPABLE and leading interdisciplinary coordination of individual beneficiary care; Intervention and implementation strategy fidelity data will be placed in a dashboard for audit and provided to IFs. IFs will use the data to provide feedback to clinicians; and develop action plans for improvement in training or care
  MiCAP with IF and EF (Main Trial): Sites will conduct MiCAP strategies described above in "MiCAP with IF" with an addition of External Facilitation. Centralized Oversight will be conducted by External Facilitators. External Facilitators will train in facilitation. The work of the External Facilitators will be tailored (i.e., type of discipline) to each site's needs. Intervention and implementation strategy fidelity data will be placed in a dashboard and will be provided to External Facilitators. External Facilitators will use the data to provide feedback to Internal Facilitators; and develop action plans for improvement in site clinician training or beneficiary care as needed.
Arm/Group | MiCAP With IF (Main Trial) | MiCAP With IF and EF (Main Trial)
Number analyzed (Participants) | 282 | 257
Score on scale | -2.34 (0.21) | -2.57 (0.30)
Statistical Analysis 1: Comparison: MiCAP With IF (Main Trial) vs MiCAP With IF and EF (Main Trial); Test type: Other — Examination of clinician self-efficacy on facilitation (IF vs IF+EF) (baseline to exit) when using an evidence-based intervention (CAPABLE); p = 0.54, Mixed Models Analysis — Threshold for statistical significance was .05 with no adjustments for multiple testing; Nesting of clinicians within site was adjusted for as a random effect; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.51 to 0.97], Standard Error of Mean 0.36

11. Other Pre Specified Outcome: Administrative Supplement: Feasibility of Use of Intervention With Clinicians, Caregivers and Beneficiaries.
Description: Feasibility of use of intervention with caregivers use of toolkit with beneficiaries with Alzheimer's Disease or dementia following implementation of CAPABLE.
  Feasibility was measured as: the percentage of those who consented and enrolled of those who were recruited who were eligible.
Time Frame: Recruitment period of 9-months.
Population: Caregivers: >21 years of age, an Informal Caregiver for a beneficiary in Medicaid waiver program.
  Clinicians: >21 years of age employed as RN or SW in waiver program where study conducted.
  Beneficiary: >21 years of age and enrolled in waiver program, and diagnosed with Alzheimer's disease or other dementia.
  NOTES:
  * 1 Overall Number of Participants Analyzed: is the total number recruited.
  * 2 The Measure Type in Outcome Measure Data Table is the number enrolled of the number recruited.
Measure: Count of Participants; unit: Participants
Groups:
- Administrative Supplement: Caregivers: Caregivers enrolled in trial to assist with providing CAPABLE to beneficiaries.
- Clinicians Enrolled in Study.: Clinicians employed at waiver sites that worked with caregivers and cared for beneficiaries.
- Beneficiaries Enrolled in the Study.: A waiver participant who has an informal caregiver and a diagnosis of Alzheimer's disease or dementia.
Arm/Group | Administrative Supplement: Caregivers | Clinicians Enrolled in Study. | Beneficiaries Enrolled in the Study.
Number analyzed (Participants) | 58 | 135 | 60
Participants | 50 | 106 | 52

12. Other Pre Specified Outcome: Administrative Supplement: Acceptability of Caregiver Use of Intervention With Beneficiaries.
Description: Acceptability of Caregiver Use of Toolkit With Beneficiaries With Alzheimer's Disease or Dementia Following Implementation of CAPABLE. Acceptability: counts of toolkit use and sections used.
Time Frame: 9-months
Population: Informal caregivers enrolled in study to care for beneficiaries in the waiver program.
Measure: Number; unit: Count of caregiver use of toolkit
Groups:
- Administrative Supplement: Group-Caregivers: Caregivers enrolled in study to care for beneficiaries in the waiver program.
Arm/Group | Administrative Supplement: Group-Caregivers
Number analyzed (Participants) | 50
Count of caregiver use of toolkit | 813

13. Other Pre Specified Outcome: Administrative Supplement: Beneficiaries Outcomes Activities of Daily Living (ADL), Instrumental Activities of Daily Living (IADLs), Pain and Depression) Pre-/Post-intervention From Minimum Data Set-Home Care MDS-HC.
Description: Activities of Daily Living: 11 items each rated as 0=Independent, 1=Set-up help, 2=Supervision, 3=Limited assist, 4=Extensive assist, 5=Maximal assist, 6=Total dependence; summed score ranged 0-66; higher score=worse Activities of Daily Living
  Instrumental Activities of Daily Living: 8 items each rated as 0=Independent, 1=Set-up help, 2=Supervision, 3=Limited assist, 4 Extensive assist, 5=Maximal assist, 6=Total dependence; summed score ranged 0-48; higher score=worse Instrumental Activities of Daily Living
  Pain: 4 items; ranges for frequency 0-3, intensity 0-4, consistency 0-3, breakthrough 0-1; summed score ranged 0-11; lower score=less pain.
  Depression: 3 items little interest in things; anxious, restless, or uneasy; and sad, depressed, or hopeless; scored as 0=Not in last 3 days, 1=Not in last 3 days, but often feels that way, 2=In 1-2 days of last 3 days, 3=Daily in last 3 days, 8=Person could/would not respond; summed score ranged 0-24; lower score=less depressed
Time Frame: Baseline (0-months) compared to Exit (9-months)
Population: Beneficiaries with Alzheimer's Disease or other dementia in the waiver program.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Administrative Supplement: Beneficiaries Baseline.; Administrative Supplement: Beneficiaries Exit.: Beneficiaries in waiver program with Alzheimer's Disease or dementia.
Arm/Group | Administrative Supplement: Beneficiaries Baseline. | Administrative Supplement: Beneficiaries Exit.
Number analyzed (Participants) | 52 | 52
Score on scale
  Depression | 5.52 (8.75) | 4.52 (4.47)
  IADLs | 42.69 (9.67) | 42.22 (11.40)
  ADLs | 22.44 (17.09) | 23.49 (19.56)
  Pain | 2.85 (2.91) | 5.56 (3.36)
Statistical Analysis 1: Comparison: Administrative Supplement: Beneficiaries Baseline. vs Administrative Supplement: Beneficiaries Exit; Pain; Test type: Superiority — Pre-/post-intervention comparison; p < .01, t-test, 2 sided; Mean Difference (Net) = -2.69, 95% CI 2-sided [-3.96 to -1.42], Standard Error of Mean 1.63 — Pre minus post
Statistical Analysis 2: Comparison: Administrative Supplement: Beneficiaries Baseline. vs Administrative Supplement: Beneficiaries Exit; ADL; Test type: Superiority; p = .58, t-test, 2 sided — Threshold for statistical significance was .05 with no adjustments for multiple comparisons; Mean Difference (Net) = 1.05, 95% CI 2-sided [-2.80 to 4.91], Standard Error of Mean 1.90
Statistical Analysis 3: Comparison: Administrative Supplement: Beneficiaries Baseline. vs Administrative Supplement: Beneficiaries Exit; IADL; Test type: Superiority; p = .44, t-test, 2 sided — Threshold for statistical significance was .05 with no adjustments for multiple comparisons; Mean Difference (Net) = 1.05, 95% CI 2-sided [-2.80 to 4.91], Standard Error of Mean 1.29
Statistical Analysis 4: Comparison: Administrative Supplement: Beneficiaries Baseline. vs Administrative Supplement: Beneficiaries Exit; Depression; Test type: Superiority; p = .38, t-test, 2 sided — Threshold for statistical significance was .05 with no adjustments for multiple comparisons; Mean Difference (Net) = 1.46, 95% CI 2-sided [-1.85 to 4.77], Standard Error of Mean 1.63 — Pre minus post

14. Other Pre Specified Outcome: Administrative Supplement: Caregiver Self Efficacy and Satisfaction With Use of Intervention.
Description: Self-efficacy and satisfaction of Caregiver Use of intervention With Beneficiaries With Alzheimer's Disease or Dementia Following Implementation of CAPABLE. Efficacy effect size of intervention use on beneficiary outcomes from Parent Trial.
  SELF-EFFICACY TOOL: General Self-efficacy (GSE) is a 10-item tool (Cronbach .79-.90) with a 4-point scale summed to 0-40, with a higher score indicating more or higher self-efficacy. Cronbach's alpha at baseline was .91 for the caregiver GSE.
  SATISFACTION TOOL: Developed by PI and Team. There were 3-items measured on a scale of 1 to 10 (reported as individual concepts; not summed), with 10 being the highest satisfaction. Question 1 Content: How satisfied were you with the Toolkit content? (range 1-10). Question 2 Format: How satisfied were you with the format of the Toolkit? (range 1-10). Question 3 Helpfulness: How helpful was the Toolkit? (range 1-10)".
Time Frame: Self-efficacy: baseline (month-0) and Exit (month-4). Satisfaction: Monthly for month 0 (baseline), 1, 2, 3, 4 (exit)
Population: Informal caregivers who care for beneficiaries with Alzheimer's Disease or other dementia's in waiver program. Data not collected on the following items. Self-efficacy at Month 1, Month 2 or Month 3 (only collected at baseline month-0 and exit month-4). Satisfaction with Content of Intervention, Format of Intervention, and Helpfulness of Intervention was not collected at Baseline Month-0 (only collected at Month 1-Month-2, Month-3, Month-4 Exit).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Administrative Supplement: Group-Caregivers (Baseline Month-0); Administrative Supplement: Group-Caregivers (Exit Month-4); Administrative Supplement: Group-Caregivers (Month-1); Administrative Supplement: Group-Caregivers (Month-2); Administrative Supplement: Group-Caregivers (Month-3): Caregivers enrolled in study to care for beneficiaries in the waiver program.
Arm/Group | Administrative Supplement: Group-Caregivers (Baseline Month-0) | Administrative Supplement: Group-Caregivers (Exit Month-4) | Administrative Supplement: Group-Caregivers (Month-1) | Administrative Supplement: Group-Caregivers (Month-2) | Administrative Supplement: Group-Caregivers (Month-3)
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50
units on a scale
  Self-efficacy: number analyzed (Participants) | 50 | 50 | 0 | 0 | 0
  Self-efficacy | 2.67 (0.62) | 3.42 (0.38) |  |  |
  Satisfaction with content of intervention: number analyzed (Participants) | 0 | 50 | 50 | 50 | 50
  Satisfaction with content of intervention |  | 8.87 (1.70) | 9.03 (1.65) | 9.07 (1.44) | 8.60 (2.27)
  Satisfaction with format of intervention: number analyzed (Participants) | 0 | 50 | 50 | 50 | 50
  Satisfaction with format of intervention |  | 8.95 (1.77) | 9.58 (0.84) | 9.28 (1.25) | 9.33 (1.71)
  Helpfulness of intervention: number analyzed (Participants) | 0 | 50 | 50 | 50 | 50
  Helpfulness of intervention |  | 7.98 (2.16) | 8.79 (1.88) | 8.79 (1.88) | 8.23 (2.34)
Statistical Analysis 1: Comparison: Administrative Supplement: Group-Caregivers (Baseline Month-0) vs Administrative Supplement: Group-Caregivers (Exit Month-4); Self-efficacy change baseline (month-0) to exit (month-4); Test type: Superiority — Self-efficacy; p < 0.01, t-test, 2 sided — Threshold for statistical significance was .05 with no adjustments for multiple comparisons; Mean Difference (Net) = -0.81, 95% CI 2-sided [-1.02 to -0.60], Standard Deviation 0.11 — Pre minus post

15. Other Pre Specified Outcome: Administrative Supplement: Clinician Satisfaction With Training and Use of Intervention.
Description: Clinician satisfaction with training and use of caregiver to assist with intervention. Satisfaction: was measured using a Likert scored tool evaluating level of satisfaction (scale 1-10 with 1 being poorest).
Time Frame: 9-months
Population: There are three groups in this study: Clinicians at 3 sites who work with the caregivers to help them care for the beneficiaries in the waiver program.
Measure: Mean (Standard Deviation); unit: Satisfaction rate (scale 1-10, 1=poorest
Groups:
- Administrative Supplement: Group-Clinicians.: Clinicians who were employed at the waiver sites and were trained in using the toolkit when implementing CAPABLE with caregivers of beneficiaries with Alzheimer's Disease or Dementia.
Arm/Group | Administrative Supplement: Group-Clinicians.
Number analyzed (Participants) | 106
Satisfaction rate (scale 1-10, 1=poorest
  Satisfaction with content | 8.09 (1.60)
  Satisfaction with format | 7.55 (2.06)
  Satisfaction with newness of content for caregiver | 8.35 (1.50)
  Satisfaction with newness of content for clinician | 7.85 (1.92)
  Intent to use new information | 8.23 (1.71)
Statistical Analysis 1: Comparison: Administrative Supplement: Group-Clinicians; Test type: Other — Score on scale; p < .01, t-test, 2 sided; Mean = 8.09, Standard Deviation 1.60
Statistical Analysis 2: Comparison: Administrative Supplement: Group-Clinicians; Satisfaction with format; Test type: Other; p < .01, t-test, 2 sided; Mean = 7.55, Standard Deviation 2.06
Statistical Analysis 3: Comparison: Administrative Supplement: Group-Clinicians; Satisfaction with newness of content for caregiver; Test type: Other; p < .01, Difference from zero; Mean = 8.35, Standard Deviation 1.50
Statistical Analysis 4: Comparison: Administrative Supplement: Group-Clinicians; Satisfaction with newness of content for clinician; Test type: Other; p < .01, Difference from zero; Mean = 7.85, Standard Deviation 1.92
Statistical Analysis 5: Comparison: Administrative Supplement: Group-Clinicians; Intent to use new information; Test type: Other; p < .01, Difference from zero; Mean = 7.85, Standard Deviation 1.92

ADVERSE EVENTS:
Time Frame: Main Study: adverse event data were collected baseline through month 9. Administrative Supplement: adverse event data were collected baseline through month 4.
Arm/Group | MiCAP With IF (Main Study: Beneficiaries) | MiCAP With IF and EF (Main Study: Beneficiaries) | MiCAP With IF (Main Study: Clinicians) | MiCAP With IF and EF (Main Study: Clinicians) | Administrative Supplement: Clinicians | Administrative Supplement: Caregivers | Administrative Supplement: Beneficiaries
All-Cause Mortality (participants affected / at risk) | 0/3497 | 0/3533 | 0/282 | 0/257 | 0/106 | 0/50 | 7/52
Serious Adverse Events (participants affected / at risk) | 0/3497 | 0/3533 | 0/282 | 0/257 | 0/106 | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 0/3497 | 0/3533 | 0/282 | 0/257 | 0/106 | 0/50 | 7/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiCAP With IF (Main Study: Beneficiaries) (N=3497) | MiCAP With IF and EF (Main Study: Beneficiaries) (N=3533) | MiCAP With IF (Main Study: Clinicians) (N=282) | MiCAP With IF and EF (Main Study: Clinicians) (N=257) | Administrative Supplement: Clinicians (N=106) | Administrative Supplement: Caregivers (N=50) | Administrative Supplement: Beneficiaries (N=52)
3. Other (Not Including Serious) Adverse Events: anticipated and unanticipated events (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) — Anticipated death due to old age and aging.

LIMITATIONS AND CAVEATS:
Main Study: we were unable to collect data on fidelity to intervention (CAPABLE) use in the electronic health record during the trial as COVID Pandemic minimal documentation standards were in effect due to short staffing which limited data entry by clinicians.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (7):
  • Study Protocol and Statistical Analysis Plan: Administrative Supplement (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03634033/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Main Study (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03634033/Prot_SAP_001.pdf
  • Informed Consent Form: Main Study - Beneficiaries (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03634033/ICF_002.pdf
  • Informed Consent Form: Main Study - Clinicians (2019-02-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03634033/ICF_003.pdf
  • Informed Consent Form: Administrative Supplement - Beneficiary LAR DPOA (2021-07-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03634033/ICF_004.pdf
  • Informed Consent Form: Administrative Supplement - Caregiver (2021-07-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03634033/ICF_005.pdf
  • Informed Consent Form: Administrative Supplement - Clinician (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT03634033/ICF_006.pdf